CLINICAL TRIAL: NCT06609291
Title: Telematic Prenatal Psychological Intervention for Preventing Anxious Symptomatology
Brief Title: Anxiety is One of the Most Frequent Disorders During the Perinatal Stage Which is Associated with Adverse Health Effects for Women and Their Babies. This Study Will Be to Evaluate the Effectiveness of a Telematic Cognitive-behavioral Preventive Intervention to Manage Anxiety During Pregnancy.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Alba Val Noguerol, Principal Investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/183
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Anxiety Disorder (Panic Disorder or GAD); Anxiety Symptoms
Keywords: prevention; telematic; pregnancy; perinatal anxiety; perinatal depression
MeSH Terms: conditions — Anxiety Disorders; Panic Disorder; Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): The intervention group, who will receive the intervention protocol. The psychological intervention will consist of 7 group sessions, conducted weekly, with a duration of approximately 60 minutes each.
  Interventions: Behavioral: Telematic Prenatal Psychological Intervention for Preventing Anxious Symptomatology
- Control group (No Intervention): The control group will receive the usual care, which consists of attending follow-up and follow-up appointments for pregnancy, resolving any doubts that may arise during the process with the midwives and attending prenatal preparation classes.

INTERVENTIONS:
Behavioral: Telematic Prenatal Psychological Intervention for Preventing Anxious Symptomatology — The psychological intervention will consist of 7 group sessions, conducted weekly, with a duration of approximately 60 minutes each, with the exception of the first and last ones, which will last an hour and a half, since they will carry out the presentation and evaluation of the intervention, respectively. In turn, the program will be divided into 3 modules. Module 1. Psychoeducation and awareness about perinatal mental health, which provides information on the prevalence of anxious symptoms in the perinatal stage and the consequences for mothers and babies. Module 2. Management of emotions and thoughts. It covers 3 sessions and aims to provide strategies to identify and restructure those thoughts that harm us, as well as recognize the behaviors and emotions that they generate. Module 3. Aimed at teaching how to solve problems effec-tively and communicate in the best possible way.
  Arms: Experimental group

SUMMARY:
Anxiety is one of the most frequent disorders during the perinatal stage which is associated with adverse health effects for women and their babies. In spite of this, preventive interventions during this stage are scarce. The National Institute for Health and Clinical Excellence recommends psychological interventions, such as cognitive behavioral therapy, as a first-line treatment for mild and moderate prenatal anxiety. Early detention of anxiety symptoms in the perinatal stage can help prevent the development of more serious mental health problems. However, there are barriers to accessing interventions during this period. A long-distance intervention carried out during the pregnancy can be an effective and accessible resource to help improve women's emotional state. The primary objective of the current study is to determine whether a preventive psychological intervention developed through videoconferencing is superior to the usual care during pregnancy (attendance at pregnancy follow-up consultations and information and answers to frequently asked questions provided by the midwife) to prevent anxious symptoms during pregnancy. The secondary objective is to examine whether this same intervention is more effective than usual care in preventing depressive symptoms during pregnancy, as well as anxious and depressive symptoms in the postpartum.

A random clinical trial will be carried out among pregnant women in Spain. A recruitment of 130 participants is proposed with random assignment to one of two conditions (65 per group): (a) the experimental group will receive the cognitive-behavioral intervention via videoconference or (b) the control group will receive usual care pregnancy (attendance at pregnancy follow-up consultations and information and answers to frequently asked questions provided by the midwife).

The psychological intervention will take place via videoconference in seven weekly sessions, lasting one hour each, with groups of 6 - 8 pregnant women. A blinded assessment will be conducted through online self-administered testing at baseline, post-intervention, and at follow-up at one month, 3 and 6 months. A clinical interview will also be conducted to evaluate generalized anxiety disorder (GAD), at the same time times. Our primary hypothesis is that the intervention will decrease the frequency of women who present anxious symptomatology during pregnancy. The second objective is to analyze the effectiveness of this intervention to prevent depressive symptomatology during pregnancy, as well as postpartum anxious and depressive symptomatology.

DETAILED DESCRIPTION:
Anxiety is one of the most frequent disorders during the perinatal stage. Its prevalence is between 15% and 23% during the pregnancy, and between 3,7% and 15,0% during postpartum. In Spain, the prevalence of anxiety ranges from 16.8% to 19.5% throughout pregnancy. Additionally, one in ten women will experience comorbid anxiety and depression during pregnancy and one in twelve during the postpartum period. Although its prevalence is high, research in treating anxiety during this period is recent.

Perinatal anxiety is associated with adverse health effects for women and their babies. Regarding mothers, it has been associated to an increased probability of developing postpartum depression, a higher risk of preeclampsia, obstetric complications and bonding problems. As for newborns, they have been found to be more likely to have lower birth weight and poor cognitive development, among others. Hence the importance of detecting and intervening early in prenatal anxiety to promote the well-being of mothers and children, because despite the negative consequences associated with perinatal anxiety, the majority of women are not detected or treated, as less than 15% receive treatment. Given the high prevalence of prenatal anxiety and the potential for adverse consequences, early treatment is recommended. Evidence on the effectiveness of psychological interventions during pregnancy is scarce highlighting the importance of having specific interventions.

The National Institute for Health and Clinical Excellence recommends psychological interventions, such as cognitive behavioral therapy, as a first-line treatment for mild and moderate prenatal anxiety. Early detention of anxiety symptoms in the perinatal stage can help prevent the development of more serious mental health problems.

During pregnancy, women frequently go to health services and are more willing to receive help because they believe it will have a positive impact on their baby. However, there are barriers to accessing interventions during this period, such as lack of information about emotional problems, available and effective intervention options, as well as practical limitations of access to in-person treatment, such as costs, geographical distance, waiting lists or logistical problems such as attending appointments. Furthermore, due to the stigmatization of mental health, especially during the perinatal period, women are reluctant to attend specialized mental health clinics in person.

The advances in information and communication technologies make it possible to have interventions via the internet, which can be carried out through computers, tablets or smartphones. They have the advantage of helping to overcome the aforementioned barriers, since they improve the acceptance of the intervention, are more flexible and accessible. Systematic reviews of internet-based interventions during the perinatal period conclude that these interventions can reduce anxiety among mothers and improve depressive and anxious symptoms.

During the perinatal stage, interventions carried out through the internet represent a tool with great potential, as they tend to be more attractive, since they reduce the need to travel, one of the barriers associated with low access to treatments for psychological problems during the perinatal period. Peragallo-Urrutia et al. found that 94.0% of pregnant and postpartum women use the internet, and 83% indicate their willingness to receive an online intervention in the perinatal period.

A form of therapy applied online is teletherapy, which has gained special importance since the COVID-19 pandemic. This form of treatment is carried out following a process similar to that of face-to-face therapy, although the interaction occurs electronically. A systematic review on telepsychology showed the effectiveness of different approaches, mostly based on the cognitive behavioral model, to reduce emotional distress. However, most of the research on the prevention of perinatal anxiety through the internet is unguided interventions, where participants access an application or web platform and view the material whenever they want and do not contact with an online healthcare professional at any moment or guided, where the participants in addition to accessing the program material, have contact (via online and/or telephone) with a professional at some point during the intervention. To date, no protocol or study has been published on the effectiveness of cognitive behavioral therapy applied in a telematic format, that is, through video calls. Having an intervention developed through videoconferencing could help reduce the limitations of unguided therapies, since they do not offer a direct interaction between the therapist and the patient, nor do they address the needs that may arise during said intervention.

On the other hand, it is worth remembering the high comorbidity between anxiety and depression. In a review and meta-analysis whose objective was to evaluate the effectiveness of psychological interventions to reduce perinatal anxiety, it was found that psychological interventions aimed at reducing anxiety during the perinatal stage were also effective in reducing symptoms of depression. This supports research suggesting that transdiagnostic interventions targeting both anxious and depressive symptoms tailored to the perinatal period, may be more beneficial than disorder-specific interventions, and indicates the need to create transdiagnostic interventions to address symptoms of anxiety and depression in women during the perinatal stage, since these comorbidities are generally not recognized or treated.

The objective of this study will be to evaluate the effectiveness of a telematic cognitive-behavioral preventive intervention during pregnancy, for the management of anxiety symptoms.

After completion of the baseline questionnaire, participants will be randomly assigned to either the intervention or control group using block randomization, a 2:1 ratio, using an online randomization program. Study personnel are unaware of which treatment group each participant will be assigned to at the time of the baseline assessment.

Referring to clinical trials on psychological interventions for perinatal depression and anxiety, the power calculation was based on detecting an effect size of medium magnitude (d = 0.55) at follow-ups among participants. The investigators calculated that a sample size of 45 participants would result in a power of 0,95 with alpha set at 0,05. To guard against an expected loss to follow-up of approximately 30%, the investigators planned to enroll 65 participants in each condition.

This study is conducted according to the principles expressed in the Declaration of Helsinki and has been approved by Comité Ético de Investigación de Galicia (CEIC) of Spain. All participants are guaranteed confidentiality of the information collected throughout the process. Participation will be completely voluntary and free, and no incentive (financial or otherwise) will be received for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years of age living in the Region of Galicia (Spain)
* Pregnant with a gestational age ≤ 16
* Understand and speak Spanish fluently
* Informed consent to participate in the study
* Accessibility to the internet and a digital device ( computer, tablet or smartphone)

Exclusion Criteria:

* High-risk pregnancy or twins
* Being pharmacological treatment for anxiety and/or depression
* Not giving their consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Reduced anxiety | pre-intervention (baseline: t0), post-intervention (baseline: t1), follow-up at 1 month (t2), follow-up at 3 months (t3) and follow-up at 6 months (t4).
  The Edinburgh Depression Scale - Anxiety Subscale (EDS-3A) is the anxiety subscale of the Edinburgh Postnatal Depression Scale (EPDS). Three items (3, 4, 5) can detect anxiety in women during the perinatal period. Each of the three items has four response options (0= none, 1= somewhat, 2= quite a bit, and 3= a lot). The total score of the subscale ranges from 0 to 9. The cut-off point used in the EDS-3A to detect anxious symptomatology will be ≥ 5.
Reduced anxiety | pre-intervention (baseline: t0), post-intervention (baseline: t1), follow-up at 1 month (t2), follow-up at 3 months (t3) and follow-up at 6 months (t4).
  The State-Trait Anxiety Inventory (STAI) assesses both the current level of anxiety and the individual's predisposition to suffering from anxiety. It consists of 40 items, 20 of which refer to the state subscale (STAI-E), with the other 20 referring to the trait subscale (STAI-R). The score for each subscale ranges from 0 to 60, with higher scores indicating higher levels of anxiety. In this case, the State Anxiety Subscale (STAI-E) will be applied and the recommended cut-off point for women is greater than 31 (75th percentile).
Reduced anxiety | pre-intervention (baseline: t0), post-intervention (baseline: t1), follow-up at 1 month (t2), follow-up at 3 months (t3) and follow-up at 6 months (t4).
  Generalized Anxiety Disorder Screener (GAD-7) is a self-administered instrument consisting of 7 items with 4 response options. The total score ranges from 0 to 21, with the highest scores being the most severe. The cut-off point used to detect anxious symptoms will be ≥ 7.
Reduced generalized anxiety disorder | pre-intervention (baseline: t0), post-intervention (baseline: t1), follow-up at 1 month (t2), follow-up at 3 months (t3) and follow-up at 6 months (t4).
  The SCID is a semi-structured interview that determines formal diagnosis according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5). To diagnose generalized anxiety, you need to have had anxiety on most days in the last 6 months in at least three contexts of your daily life and show 3 of the 6 anxiety symptoms that are described in the manual. The use of such interviews improves diagnostic reliability by standardizing the assessment process and increases the diagnostic validity by facilitating the application of DSM diagnostic criteria and the systematic enquiry of symptoms that might otherwise go unnoticed.

SECONDARY OUTCOMES:
Reduced depression | pre-intervention (baseline: t0), post-intervention (baseline: t1), follow-up at 1 month (t2), follow-up at 3 months (t3) and follow-up at 6 months (t4).
  The Edinburgh Depression Scale (EPDS) is a self-reported questionnaire consisting of 10 items with 4 response options. The scores range between 0 and 30, with higher scores indicating a greater severity of depression. The Spanish validation of the EPDS for use in pregnancy will be used, and determines that the most appropriate cut-off point for screening for probable antenatal depression is 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultade de Psicoloxía, Universidade de Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
Researchers will report study results through publications.

REFERENCES:
- [Background] McCabe-Beane JE, Stasik-O'Brien SM, Segre LS. Anxiety Screening During Assessment of Emotional Distress in Mothers of Hospitalized Newborns. J Obstet Gynecol Neonatal Nurs. 2018 Jan;47(1):105-113. doi: 10.1016/j.jogn.2017.01.013. Epub 2017 May 18. PMID 28528808
- [Background] Loughnan SA, Butler C, Sie AA, Grierson AB, Chen AZ, Hobbs MJ, Joubert AE, Haskelberg H, Mahoney A, Holt C, Gemmill AW, Milgrom J, Austin MP, Andrews G, Newby JM. A randomised controlled trial of 'MUMentum postnatal': Internet-delivered cognitive behavioural therapy for anxiety and depression in postpartum women. Behav Res Ther. 2019 May;116:94-103. doi: 10.1016/j.brat.2019.03.001. Epub 2019 Mar 8. No abstract available. PMID 30877878
- [Background] Peragallo Urrutia R, Berger AA, Ivins AA, Beckham AJ, Thorp JM Jr, Nicholson WK. Internet Use and Access Among Pregnant Women via Computer and Mobile Phone: Implications for Delivery of Perinatal Care. JMIR Mhealth Uhealth. 2015 Mar 30;3(1):e25. doi: 10.2196/mhealth.3347. PMID 25835744
- [Background] Ruiz-Segovia N, Rodriguez-Munoz MF, Olivares ME, Izquierdo N, Coronado P, Le HN. Healthy Moms and Babies Preventive Psychological Intervention Application: A Study Protocol. Int J Environ Res Public Health. 2021 Nov 27;18(23):12485. doi: 10.3390/ijerph182312485. PMID 34886212
- [Background] Bayrampour H, Trieu J, Tharmaratnam T. Effectiveness of eHealth Interventions to Reduce Perinatal Anxiety: A Systematic Review and Meta-Analysis. J Clin Psychiatry. 2019 Jan 22;80(1):18r12386. doi: 10.4088/JCP.18r12386. PMID 30688418
- [Background] Loughnan SA, Joubert AE, Grierson A, Andrews G, Newby JM. Internet-delivered psychological interventions for clinical anxiety and depression in perinatal women: a systematic review and meta-analysis. Arch Womens Ment Health. 2019 Dec;22(6):737-750. doi: 10.1007/s00737-019-00961-9. Epub 2019 May 17. PMID 31101993
- [Background] Goodman JH. Women's attitudes, preferences, and perceived barriers to treatment for perinatal depression. Birth. 2009 Mar;36(1):60-9. doi: 10.1111/j.1523-536X.2008.00296.x. PMID 19278385
- [Background] Fonseca A, Canavarro MC. Women's intentions of informal and formal help-seeking for mental health problems during the perinatal period: The role of perceived encouragement from the partner. Midwifery. 2017 Jul;50:78-85. doi: 10.1016/j.midw.2017.04.001. Epub 2017 Apr 5. PMID 28395200
- [Background] Bina R, Glasser S. Factors associated with attitudes toward seeking mental health treatment postpartum. Women Health. 2019 Jan;59(1):1-12. doi: 10.1080/03630242.2017.1421286. Epub 2018 Jan 24. PMID 29281589
- [Background] Yazdanimehr R, Omidi A, Sadat Z, Akbari H. The Effect of Mindfulness-integrated Cognitive Behavior Therapy on Depression and Anxiety among Pregnant Women: a Randomized Clinical Trial. J Caring Sci. 2016 Sep 1;5(3):195-204. doi: 10.15171/jcs.2016.021. eCollection 2016 Sep. PMID 27752485
- [Background] Smith MV, Shao L, Howell H, Wang H, Poschman K, Yonkers KA. Success of mental health referral among pregnant and postpartum women with psychiatric distress. Gen Hosp Psychiatry. 2009 Mar-Apr;31(2):155-62. doi: 10.1016/j.genhosppsych.2008.10.002. Epub 2008 Dec 3. PMID 19269536
- [Background] Green SM, Donegan E, McCabe RE, Streiner DL, Agako A, Frey BN. Cognitive behavioral therapy for perinatal anxiety: A randomized controlled trial. Aust N Z J Psychiatry. 2020 Apr;54(4):423-432. doi: 10.1177/0004867419898528. Epub 2020 Jan 20. PMID 31957479
- [Background] Sanchez SE, Puente GC, Atencio G, Qiu C, Yanez D, Gelaye B, Williams MA. Risk of spontaneous preterm birth in relation to maternal depressive, anxiety, and stress symptoms. J Reprod Med. 2013 Jan-Feb;58(1-2):25-33. PMID 23447915
- [Background] Ding XX, Wu YL, Xu SJ, Zhu RP, Jia XM, Zhang SF, Huang K, Zhu P, Hao JH, Tao FB. Maternal anxiety during pregnancy and adverse birth outcomes: a systematic review and meta-analysis of prospective cohort studies. J Affect Disord. 2014 Apr;159:103-10. doi: 10.1016/j.jad.2014.02.027. Epub 2014 Feb 26. PMID 24679397
- [Background] Field T. Prenatal anxiety effects: A review. Infant Behav Dev. 2017 Nov;49:120-128. doi: 10.1016/j.infbeh.2017.08.008. Epub 2017 Sep 5. PMID 28886563
- [Background] Farre-Sender B, Torres A, Gelabert E, Andres S, Roca A, Lasheras G, Valdes M, Garcia-Esteve L. Mother-infant bonding in the postpartum period: assessment of the impact of pre-delivery factors in a clinical sample. Arch Womens Ment Health. 2018 Jun;21(3):287-297. doi: 10.1007/s00737-017-0785-y. Epub 2017 Oct 18. PMID 29046965
- [Background] Alipour Z, Lamyian M, Hajizadeh E. Anxiety and fear of childbirth as predictors of postnatal depression in nulliparous women. Women Birth. 2012 Sep;25(3):e37-43. doi: 10.1016/j.wombi.2011.09.002. Epub 2011 Sep 29. PMID 21959041
- [Background] Loughnan SA, Wallace M, Joubert AE, Haskelberg H, Andrews G, Newby JM. A systematic review of psychological treatments for clinical anxiety during the perinatal period. Arch Womens Ment Health. 2018 Oct;21(5):481-490. doi: 10.1007/s00737-018-0812-7. Epub 2018 Jan 24. PMID 29368048
- [Background] Clinkscales N, Golds L, Berlouis K, MacBeth A. The effectiveness of psychological interventions for anxiety in the perinatal period: A systematic review and meta-analysis. Psychol Psychother. 2023 Jun;96(2):296-327. doi: 10.1111/papt.12441. Epub 2022 Dec 11. PMID 36504355
- [Background] Falah-Hassani K, Shiri R, Dennis CL. The prevalence of antenatal and postnatal co-morbid anxiety and depression: a meta-analysis. Psychol Med. 2017 Sep;47(12):2041-2053. doi: 10.1017/S0033291717000617. Epub 2017 Apr 17. PMID 28414017
- [Background] Val A, Miguez MC. Prevalence of Antenatal Anxiety in European Women: A Literature Review. Int J Environ Res Public Health. 2023 Jan 8;20(2):1098. doi: 10.3390/ijerph20021098. PMID 36673854
- [Background] Sinesi A, Maxwell M, O'Carroll R, Cheyne H. Anxiety scales used in pregnancy: systematic review. BJPsych Open. 2019 Jan;5(1):e5. doi: 10.1192/bjo.2018.75. PMID 30762504
- [Background] Dennis CL, Falah-Hassani K, Shiri R. Prevalence of antenatal and postnatal anxiety: systematic review and meta-analysis. Br J Psychiatry. 2017 May;210(5):315-323. doi: 10.1192/bjp.bp.116.187179. Epub 2017 Mar 16. PMID 28302701